CLINICAL TRIAL: NCT02660112
Title: A Phase II, Open Label Prospective Single Center Drug Study Evaluating the Safety and Efficacy of (+)-Epicatechin in Subjects With Friedreich's Ataxia
Brief Title: (+) Epicatechin to Treat Friedreich's Ataxia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ralitza Gavrilova (Other)
Collaborators: Cardero Therapeutics, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Ralitza Gavrilova, MD, Sponsor-Investigator, Mayo Clinic
Organization: Mayo Clinic (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15-006845
Record Dates: First submitted 2016-01-18; First posted 2016-01-21 (Estimated); Results first posted 2019-12-05 (Actual); Last update posted 2019-12-05 (Actual); Status verified 2019-02

CONDITIONS: Friedreich's Ataxia
MeSH Terms: conditions — Friedreich Ataxia | interventions — Catechin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- (+)-Epicatechin (Experimental): Total daily dose 75mg (+)-Epicatechin; 25mg cap three times per day by mouth for 24 weeks
  Interventions: Drug: (+)-Epicatechin

INTERVENTIONS:
Drug: (+)-Epicatechin — 25mg (+)-Epicatechin capsules. Starting dose 75mg total daily dose (one 25mg cap taken three times per day). Dose escalation at 12 weeks for non-responders to 150mg total daily dose (two 25mg caps taken three times per day)

SUMMARY:
This 24-week study will test the safety and effectiveness of synthetically produced (+) Epicatechin in treating patients who have Friedreich's Ataxia, a neurological disorder.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of Friedreich's Ataxia (FA) by Frataxin genetic testing and/or Frataxin enzyme analysis
* Between age 10 and 50 years of age, inclusive
* Body weight of 25 kilograms or higher
* Minimum of one affected organ (cardiac or neurological) system, as evidenced by clinical signs/symptoms
* Disease duration ≤7 years, based on onset date of FA symptoms
* Has no known contraindication to gadolinium contrast such as severe allergy or Glomerular Filtration Rate <30 ml/min/m^2.
* Has no known contraindication to non-contrast Magnetic Resonance Imaging (MRI) evaluation such as pacemaker or magnetically active metal fragments.
* Women of childbearing age must:

  * Have a negative pregnancy human chorionic gonadotropin test prior to receiving study drug.
  * Agree to use contraception for the duration of the study drug dosing, plus 1 month after completion of the study.

Exclusion Criteria:

* Advanced cardiac failure, New York Heart Association (NYHA) Classification Scale-Class IV (advanced stage heart failure)
* Clinically significant comorbidities that may also lead to cardiomyopathy, for example long standing hypertension, familial cardiomyopathy.
* Clinically significant comorbidities that would, in the opinion of the investigators, compromise the interpretation of test results.
* Pregnant, breast-feeding or planning to become pregnant during study timeframe.
* Patients with contraindications to regadenoson, i. e. second- or third-degree atrioventricular (AV) block or sinus node dysfunction. Has received an investigational drug within thirty (30) days of baseline visit.
* Thrombocytopenia (<125 x 10^9/Liter) or prolonged Prothrombin Time/Partial Thromboplastin Time (PT/PTT) at baseline.
* Clinically significant hypotension (systolic blood pressure <90) due to heart failure or other conditions.

Ages: 10 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Actual)
Dates: Start 2016-09; Primary Completion 2018-12-30 (Actual); Study Completion 2018-12-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ralitza H Gavrilova, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Qureshi MY, Patterson MC, Clark V, Johnson JN, Moutvic MA, Driscoll SW, Kemppainen JL, Huston J 3rd, Anderson JR, Badley AD, Tebben PJ, Wackel P, Oglesbee D, Glockner J, Schreiner G, Dugar S, Touchette JC, Gavrilova RH. Safety and efficacy of (+)-epicatechin in subjects with Friedreich's ataxia: A phase II, open-label, prospective study. J Inherit Metab Dis. 2021 Mar;44(2):502-514. doi: 10.1002/jimd.12285. Epub 2020 Aug 31. PMID 32677106

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | (+)-Epicatechin
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | (+)-Epicatechin
Number analyzed (Participants) | 10
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 14.5 [10 to 50]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 6
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Friedreich Ataxia Rating Scale (FARS) Composite Score
Description: The Friedreich Ataxia Rating Scale (FARS) is made up of a measure of ataxia, an activities of daily living subscale and a neurological subscale. This scale also includes the 8m walk at maximum speed (8MW), the 9-hole peg test (9HPT), PATA rate (assesses speech speed by repetitions of pronouncing "PaTa" ) and low-contrast letter acuity.
  FARS is made up of a measure of ataxia, an activities of daily living subscale and a neurological subscale. This scale also includes the 8m walk at maximum speed (8MW), the 9-hole peg test (9HPT), PATA rate and low-contrast letter acuity. The scores from the three subscales are added to generate a total score ranging from 0 to 159, with a higher score indicating a greater level of disability.
Time Frame: Baseline, 24 weeks
Population: One subject did not complete week 24 questionnaire
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | (+)-Epicatechin
Number analyzed (Participants) | 9
score on a scale | 55.0 (18.72)
Statistical Analysis 1: Comparison: (+)-Epicatechin; Test type: Superiority; p = 0.336, Wilcoxon (Mann-Whitney)

2. Primary Outcome: Change in Ventricular Hypertrophy as Shown on Cardiac MRI
Description: Left ventricular mass and left ventricular (LV) mass indexed to body surface area estimated by Left Ventricle (LV)cavity dimension and wall thickness at end-diastole. Normal values of LV mass indexed to body surface area are found to be 49-115 gL/m2 in men and 43-95 g/m2 in women.
Time Frame: Baseline, 24 weeks
Measure: Mean (Standard Deviation); unit: mL/m2
Arm/Group | (+)-Epicatechin
Number analyzed (Participants) | 10
mL/m2 | 55.9 (9.49)

ADVERSE EVENTS:
Time Frame: Adverse Events were collected over a 24 week time period
Arm/Group | (+)-Epicatechin
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 3/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | (+)-Epicatechin (N=10)
Transient worsening of migraine (Nervous system disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-01-27): https://cdn.clinicaltrials.gov/large-docs/12/NCT02660112/Prot_SAP_000.pdf